CLINICAL TRIAL: NCT00235651
Title: Pharmacokinetic and Deposition Profiles of Inhaled Lipid Complex Amphotericin B (Abelcet®) in Lung Transplant Recipients (Radiotagging Protocol)
Brief Title: Abelcet Radiotagging Protocol: Inhaled Lipid Complex Abelcet® in Lung Transplant Recipients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: study completed
Sponsor: University of Pittsburgh (Other)
Collaborators: Enzon Pharmaceuticals, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB# 0509013
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Last update posted 2008-12-17 (Estimated); Status verified 2008-12

CONDITIONS: Lung Transplantation; Lung Diseases
Keywords: Lung transplant recipient
MeSH Terms: conditions — Lung Diseases | interventions — Amphotericin B

INTERVENTIONS:
Drug: Amphotericin B

SUMMARY:
The purpose of this study is to quantify the dose of aerosol medication deposited in the lungs of lung transplant recipients receiving a single nebulized treatment of aerosolized Abelcet® (lipid complexed amphotericin-B). This study is being performed to determine the range of deposited doses and patterns of distribution that could be expected in this population so that the ultimate efficacy of this preparation can be evaluated. A radioisotope technique will be utilized to track the medication dose. The study will include 12 subjects who will perform one testing session lasting approximately 3 hours. An Investigational New Drug Application (IND) detailing this protocol has been submitted by the principal investigator (PI) and approved by the Food and Drug Administration [FDA] (72,521).

DETAILED DESCRIPTION:
Research Methods:

The patient will need to complete one visit that will take about 3 hours of their time. All testing will be performed in the Nuclear Medicine Department located on the first floor of the Presbyterian Hospital.

Screening:

1. For women who could possibly be pregnant, a small amount of urine will be used for pregnancy testing to be performed on the study day prior to any drug delivery. Pregnant women, or women who are currently breast-feeding an infant, will not be allowed to take part in this study.
2. Patients will be asked a few questions that will not take more than five minutes by one of the investigators or study coordinator. These questions include information about past medical history, surgical dates, medications, etc. The patient's medical record will be reviewed for demographic information (age, sex, and race), lab results (standard post transplant care), medication information, as well as any testing/procedures that they have undergone.

Experimental Procedures:

1. Fifteen minutes prior to the administration of radiolabeled Abelcet® by nebulizer, we will measure and assess blood pressure and heart rate, assess lung sounds, perform pulmonary function testing, and re-verify that the subject has no known allergies or previous adverse experiences with radiopharmaceuticals. Female subjects will receive a urine pregnancy test on the day of testing, prior to drug administration.
2. Subjects will be seated between the heads of a dual-head gamma camera so that the region from the top of the head to the stomach is viewable by this device which depicts radioactivity inside of the body. Subjects will then inhale the test aerosol. The aerosol will be delivered using an Aeroeclipse breath actuated Nebulizer driven by a DeVilbiss 8650D compressor set to 40psig. The anterior head of the gamma camera will be moved away from the subject during aerosol administration, but imaging will be performed through the posterior head throughout the drug delivery. Drug delivery will take approximately 25 minutes.
3. When the nebulized dose has been completely delivered the nebulizer and associated equipment will be removed from the room, and the anterior head of the gamma camera will be brought back into close proximity to the subject. A series of 30s images will be taken depicting the drug deposited in the subjects. The first 4 images will be taken manually at high-pixel resolution. The camera will then be set to automatically acquire images for the next 20 minutes at lower resolution.
4. Radioactivity will be used as an analog for drug dose. The starting dose of radioactivity added to the nebulizer will be compared to the dose found in the nebulizer and exhalation filters after dose delivery, in order to determine the total dose deposited. The regional breakdown of the deposited dose will be determined using the gamma camera images.
5. While the camera heads are still in close proximity to the subject, a small amount of Xenon [Xe-133] gas will be administered to the subjects via mask so that the shape of the lungs can be depicted and imaged. This gas will then be washed out through an absorbent filter. The gas inhalation will take approximately 6 minutes.
6. After the completion of imaging (approximately 30 minutes after drug administration) subjects will be moved to a small exam room where again blood pressure, heart rate, and lung sounds will be reassessed. Pulmonary function tests will be re-performed and the change in forced expiratory volume in 1 second [FEV1] (if any) caused by the drug will be determined. Subjects will be treated with bronchodilators if exam reveals any signs of bronchoconstriction resulting from the aerosol. In addition, adverse events will be monitored and recorded.

Monitoring/Follow Up:

Each participant will undergo the following monitoring procedures to evaluate the effectiveness and safety of the experimental procedures that are not part of standard medical care.

1. The monitoring/follow-up procedures include a follow-up phone call from the study coordinator to check for any side effects of the experimental procedure. This call will take place the day after the participant has completed the experimental procedure. This call will take no longer than 5-10 minutes to complete.
2. Thirty days after participants have completed the experimental procedure, the study coordinator will call the participant to check for any side effects associated with the experimental procedure. This call will take no longer than 5-10 minutes to complete.

After this phone call the patient will have completed the study.

Rationale for Follow-Up:

The half-life of the radiopharmaceutical [Technetium (Tc-99m)] used for labeling of the drug is 6.02 hours. The serum half-life for amphotericin after intravenous (IV) Abelcet administration is of the order of 170 hours (Abelcet label). Detectable concentrations of Amphotericin have been found in the BAL fluid of the lungs after 192 hours post administration of inhaled Abelcet in our previous studies. The longer half-life associated with the active medication necessitates the longer follow up period.

ELIGIBILITY:
Inclusion Criteria:

1. Single or double lung transplant recipients
2. Age > 18
3. Willing to be available at the testing center
4. Able to understand and complete informed consent

Exclusion Criteria:

1. Pregnant women, or women capable of bearing children who will not perform urine pregnancy test.
2. Nursing mothers.
3. Hypersensitivity to amphotericin B (Abelcet®) or technetium [Tc-99m] based radiopharmaceuticals.
4. Subjects with a past history of bronchospasm associated with aerosol drug use
5. Subjects with active bacterial or viral infection as defined by the current use of non-prophylactic antibiotic anti-viral medications
6. Subjects with an FEV1 < 30% predicted or forced vital capacity (FVC) % predicted < 30%
7. Subjects requiring supplemental oxygen
8. Receipt of inhalational or IV amphotericin B within last 30 days
9. Subjects with known fungal infection, as per Mycoses Study Group (MSG) criteria, on therapy with antifungal drugs or diagnosed on the day of bronchoscopy
10. Serum creatinine > 1.9 mg/dl on the day of clinic visit
11. Liver enzymes ALT/AST/alk phos greater than two times the normal limit
12. Concurrent intravenous aminoglycoside use
13. Subjects with fever > 38.2°C
14. Subjects on mechanical ventilation.
15. Have participated in any studies involving radiopharmaceuticals within 14 days.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12
Dates: Start 2005-10; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
to determine the dose of medication deposited in the lungs

SECONDARY OUTCOMES:
to determine the regional distribution of the drug in the lungs

CONTACTS AND LOCATIONS:
Overall Officials: Shahid Husain, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States